CLINICAL TRIAL: NCT07372430
Title: Proximal Versus Distal Superior Cluneal Nerve Block in Superior Cluneal Nerve Entrapment: A Prospective, Randomized, Single-Blind Trial
Brief Title: Proximal Versus Distal Superior Cluneal Nerve Block in Entrapment Neuropathy
Status: Recruiting | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1496
Record Dates: First submitted 2026-01-06; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cluneal Syndrome
Keywords: Neuralgia; Peripheral Nerve Entrapment; low back pain
MeSH Terms: conditions — Neuralgia; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Proximal SCN Injection (Ultrasound-Guided): Ultrasound-guided proximal interfascial (plane block) approach for suspected superior cluneal nerve entrapment.
  Interventions: Procedure: Ultrasound-guided proximal superior cluneal nerve injection
- Distal SCN Injection (Ultrasound-Guided): Ultrasound-guided distal perineural approach for suspected superior cluneal nerve entrapment.
  Interventions: Procedure: Ultrasound-guided distal superior cluneal nerve injection

INTERVENTIONS:
Procedure: Ultrasound-guided distal superior cluneal nerve injection — The ultrasound probe will be placed over the posterior superior iliac crest to visualize the fibro-osseous tunnel where the superior cluneal nerve passes. Using an in-plane approach, the needle will be advanced toward the target area, and the injection will be administered at the fascial exit point of the nerve. A total injectate volume of 5 cc (2 cc bupivacaine, 2 cc dexamethasone, and 1 cc normal saline) will be administered. All procedures will be performed in the prone position under standard aseptic conditions.
  Groups: Distal SCN Injection (Ultrasound-Guided)
Procedure: Ultrasound-guided proximal superior cluneal nerve injection — Patients randomized to the proximal injection group will undergo ultrasound-guided injection above the iliac crest level. The target will be the plane beneath the posterior layer of the thoracolumbar fascia. Using an in-plane approach, the injectate will be delivered into the interfascial plane. A total injectate volume of 5 cc (2 cc bupivacaine, 2 cc dexamethasone, and 1 cc normal saline) will be administered under ultrasound guidance. Patient positioning and aseptic conditions will be identical to those used in the distal perineural injection group.
  Groups: Proximal SCN Injection (Ultrasound-Guided)

SUMMARY:
Superior cluneal nerve (SCN) entrapment is an underdiagnosed cause of chronic low back and gluteal pain. Although diagnostic nerve block is considered the gold standard for confirming SCN entrapment, there is no consensus regarding the optimal injection approach. This prospective observational study aims to compare the clinical effectiveness of proximal and distal ultrasound-guided SCN block techniques in patients diagnosed with SCN entrapment. Pain intensity and functional outcomes will be evaluated over the follow-up period to assess differences between the two approaches.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the effects of two different ultrasound-guided injection techniques on pain intensity, functional status, neuropathic pain components, and quality of life in patients with suspected superior cluneal nerve (SCN) entrapment. Pain severity will be assessed using the Visual Analog Scale (VAS), functional status using the Oswestry Disability Index (ODI), neuropathic pain components using the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS), and quality of life using the Short Form-12 (SF-12). The study aims to determine which injection technique provides superior clinical outcomes.

The secondary objective is to evaluate lumbosacral angle, lumbar lordosis angle, pelvic tilt, sacral tilt, and the presence of scoliosis, and to investigate the relationship between these postural and radiological parameters, SCN entrapment, and treatment response.

Through this study, ultrasound-guided injection techniques used in the diagnosis and treatment of SCN entrapment will be comparatively evaluated, addressing an important gap in the current literature and providing high-level scientific evidence to guide clinicians in the management of chronic low back and gluteal pain.

This study is designed as a prospective, randomized, single-blind clinical study comparing two different ultrasound-guided injection techniques in patients with suspected superior cluneal nerve entrapment. The study population will consist of patients presenting to the Algology Outpatient Clinic of Health Sciences University Gaziosmanpaşa Physical Medicine and Rehabilitation Training and Research Hospital during the study period, who meet the inclusion and exclusion criteria, have chronic low back and/or gluteal pain, are suspected of having SCN entrapment based on clinical examination, have not benefited from conservative treatment, and voluntarily agree to participate in the study.

Based on a power analysis with 95% power, a total of 54 patients are planned to be included in the study, with 27 patients allocated to each group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Chronic low back and/or gluteal pain lasting longer than 3 months
* Localized point tenderness and/or paresthesia on palpation over the unilateral posterior iliac crest
* Clinical suspicion of superior cluneal nerve entrapment based on physical examination
* Failure to respond to conservative treatment
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Active local or systemic infection
* Cognitive impairment or psychiatric disorders interfering with study participation
* History of malignancy or cancer-related pain
* Uncontrolled diabetes mellitus or severe comorbid conditions adversely affecting general health
* Pregnancy
* Known allergy to the medications used in the injection
* Prominent radicular pain associated with neurological deficit
* History of interventional procedures applied to the lumbar region within the last 6 months
* Initiation of another lumbar interventional or medical treatment during the follow-up period
* Suspected bilateral superior cluneal nerve entrapment
* Sphincter dysfunction related to neurological disease
* Bleeding diathesis or coagulation disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients aged 18 to 75 years presenting with chronic low back and/or gluteal pain lasting longer than three months, who are clinically suspected of having superior cluneal nerve entrapment based on physical examination findings. Eligible participants will be those who have not responded to conservative treatment and who attend the Algology Outpatient Clinic during the study period. Only patients with unilateral symptoms who meet all inclusion and exclusion criteria and who provide written informed consent will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, 1 month, and 3 months
  Primary Outcome Measure Visual Analog Scale for Pain (VAS): Change in pain intensity assessed using the Visual Analog Scale (VAS).The VAS is a 10-cm horizontal scale ranging from 0 (no pain) to 10 (worst imaginable pain).Higher scores indicate greater pain intensity, and a reduction in VAS score represents clinical improvement.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline, 1 month, and 3 months
  Oswestry Disability Index (ODI): Change in disability related to low back pain assessed using the Oswestry Disability Index (ODI).The validated and reliability-tested Turkish version of the ODI will be used in this study.The ODI consists of 10 items, each scored from 0 to 5, yielding a maximum total raw score of 50.The total score is converted to a percentage using the following formula:ODI percentage = (Total score / 50) × 100
  Higher percentage scores indicate greater disability. Disability levels are interpreted as follows:
  * 0-20%: Minimal disability
  * 21-40%: Moderate disability
  * 41-60%: Severe disability
  * 61-80%: Crippling disability
  * 81-100%: Bed-bound or exaggerated symptoms
  A decrease in ODI percentage score indicates improvement in functional status.
Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) | Baseline, 1 month, and 3 months
  Assessment of neuropathic pain features using the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) questionnaire.The LANSS scale consists of 7 items with a total score ranging from 0 to 24.A score of ≥12 indicates the presence of neuropathic pain mechanisms.Higher scores reflect greater neuropathic pain components.
Short Form-12 Health Survey (SF-12) | Baseline, 1 month, and 3 months
  Health-related quality of life assessed using the Short Form-12 Health Survey (SF-12).The SF-12 generates two composite scores:
  * Physical Component Summary (PCS)
  * Mental Component Summary (MCS) Both PCS and MCS scores are calculated according to standard scoring algorithms.Higher scores indicate better physical and mental health-related quality of life, respectively.In this study, PCS and MCS scores will be analyzed separately to evaluate physical and mental aspects of quality of life.
Baseline Postural and Radiological Characteristics in Patients with Superior Cluneal Nerve Entrapment | Baseline (pre-intervention)
  Baseline postural and radiological characteristics will be assessed prior to intervention in patients with superior cluneal nerve entrapment. Previously obtained standing lateral lumbosacral and pelvic radiographs will be used. Lumbar lordosis, sacral slope, lumbosacral angle, and pelvic tilt will be measured as radiographic angles in degrees on standing lateral images and categorized as decreased/normal/increased (lumbar lordosis, sacral slope, lumbosacral angle) or anterior/normal/posterior (pelvic tilt). Scoliosis will be evaluated based on physical examination and review of existing radiographs and MRI scans; when clinically indicated, standing scoliosis radiographs will be obtained. Scoliosis will be assessed using the Cobb method and recorded as present or absent. These findings will be descriptively reported.

CONTACTS AND LOCATIONS:
Overall Officials: Tugce Yavuz Mollavelioglu, MD, Study Chair — Gaziosmanapasa Educational and Training Hospital
Locations (1):
- Health Sciences University Gaziosmanpaşa Physical Medicine and Rehabilitation Training and Research Hospita, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional data protection policies and the absence of participant consent for data sharing beyond the scope of the current study.

REFERENCES:
- [Background] Nielsen TD, Moriggl B, Barckman J, et al. Randomized trial of ultrasound-guided superior cluneal nerve block. Reg Anesth Pain Med Epub. 2019;44(8):772-780. doi:10.1136/rapm-2018-100174
- [Background] Bodner G, Platzgummer H, Meng S, Bruve muayeneer GM, Lieba-Samal D. Successful identification and assessment of the superior cluneal nerves with high-resolution sonography. Pain Physician. 2016;19(3):197-202.